CLINICAL TRIAL: NCT06608667
Title: The Evaluation of Ischemia-reperfusion Injury in the Donor Liver Can Be Achieved Through the Utilization of Noninvasive Near-infrared Hyperspectral Imaging.
Brief Title: The Clinical Study Aims to Assess the Quality of Donor Livers Using Hyperspectral Imaging.
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Hu Liangshuo, Principal Investigator, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XJTU1AF2021LSK-272
Record Dates: First submitted 2024-06-11; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Liver Transplantation; Hyperspectral Imaging
Keywords: liver transplantation; Hyperspectral Imaging; Evaluation of donor liver; Early Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mild ischemia reperfusion injury group(MIRIG): Suzuki's score of 0 to 2 group were divided into mild ischemia-reperfusion injury group. Subjects matching the characteristics of this group were screened according to inclusion and exclusion criteria, and preoperative and postoperative characteristics of the corresponding recipients and donors were collected and recorded for subsequent analysis.
  Interventions: Device: The study was retrospective and did not involve the application of interventions
- Severe ischemia reperfusion injury group(SIRIG): Suzuki's score of 3 to 4 group were divided into severe ischemia-reperfusion injury group. Subjects matching the characteristics of this group were screened according to inclusion and exclusion criteria, and preoperative and postoperative characteristics of the corresponding recipients and donors were collected and recorded for subsequent analysis.
  Interventions: Device: The study was retrospective and did not involve the application of interventions

INTERVENTIONS:
Device: The study was retrospective and did not involve the application of interventions — The study was retrospective and did not involve the application of interventions

SUMMARY:
Based on hyperspectral imaging equipment, this project collected hyperspectral imaging data of donor livers, analyzed various parameters, investigated the detection capability of hyperspectral imaging for assessing donor liver quality, gathered patient prognosis information, examined the correlation between early postoperative complications and hyperspectral imaging data, and explored characteristic parameters for evaluating donor liver quality using hyperspectral imaging technology. The occurrence of early complications was predicted.

DETAILED DESCRIPTION:
Hyperspectral imaging (HSI) is an advanced optical technology that combines spectroscopy and imaging, providing a non-destructive approach for clinical diagnosis. In recent years, hyperspectral imaging has emerged as a prominent research topic in the field of applied medicine. Liver transplantation is considered the most effective treatment for end-stage liver disease; however, the scarcity of donor livers and the growing number of patients awaiting transplantation pose significant challenges to global organ transplantation. The evaluation of donor livers has always been a focal point in liver transplantation. Currently, clinical evaluation relies heavily on subjective judgment by transplant physicians based on general appearance and touch assessments, along with clinical examinations and pathological biopsy results. Nevertheless, studies have demonstrated that these methods are not entirely reliable for assessing liver quality. Therefore, it is crucial to identify additional evaluation parameters and establish a convenient, reliable, and non-invasive method to assess donor liver quality. This study aims to analyze hyperspectral imaging data alongside clinical test data and recipient complications occurring between June 2022 to June 2024 to evaluate the quality of donor livers using hyperspectral imaging technology while exploring potential evaluation parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients ranged in age from 18 to 65
2. Donor age ≥ 18 years

Exclusion Criteria:

1. Recipients are younger than 18 years or older than 65 years
2. Donor younger than 18 years
3. Secondary liver transplantation.
4. Multiple organ transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age from 18 to 65) who underwent liver transplantation using grafts from deceased donors from June 1st, 2022 to June 30st, 2024, were retrospectively identified using Chian Liver Transplant Registry(CLTR)
  , a database and official website for national data gathering and clinical data from the First Affiliated Hospital of Xi'an Jiaotong University
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Hyperspectral imaging to assess ischemia-reperfusion injury in liver grafts | From June 1,2022 to June 30,2024
  Assessment of severity of ischemia-reperfusion injury of donor liver grafts by hyperspectral imaging

SECONDARY OUTCOMES:
Assessment of fatty liver graft using hyperspectral imaging | From June 1,2022 to June 30,2024
  Assessing the severity of fatty liver using Hyperspectral Imaging
Hyperspectral imaging predicts early serologic markers of liver function and inflammatory factors | From June 1,2022 to June 30,2024
Assessing early allograft dysfunction after liver transplantation using hyperspectral imaging | From June 1,2022 to June 30,2024

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, MD PhD, Study Chair — First Affiliated Hospital Xian Jiaotong University
Locations (1):
- First Affiliated Hospital Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
The study was based on database from The First Affiliated Hospital of Xian Jiao Tong University , researchers did not have access to patients information or raw data unless approved by the Ethics Committee of The First Affiliated Hospital of Xian Jiao Tong University.